CLINICAL TRIAL: NCT00728091
Title: A Double-Blind, Randomized, Placebo-Controlled Multicenter Study Evaluating the Efficacy and Safety of Two Doses of Satavaptan (SR121463B) Versus Placebo in Patients With Dilutional Hyponatremia Due to the Syndrome of Inappropriate Antidiuretic Hormone Secretion (SIADH)
Brief Title: A Phase III Study Evaluating the Efficacy and Safety of Satavaptan Versus Placebo in Patients With Dilutional Hyponatremia
Acronym: AQUARIST1
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC10102; EudraCT:2007-007941-10
Record Dates: First submitted 2008-07-31; First posted 2008-08-05 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-04

CONDITIONS: Hyponatremia; Inappropriate ADH Syndrome
Keywords: aquaretic; SIADH
MeSH Terms: conditions — Hyponatremia; Inappropriate ADH Syndrome | interventions — satavaptan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Satavaptan Dose 1 (Experimental): Fixed Low dose up to day 4, followed by optional titration up to day 30
  Interventions: Drug: Satavaptan
- Satavaptan Dose 2 (Experimental): Fixed High dose up to day 4, followed by optional titration up to day 30
  Interventions: Drug: Satavaptan
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Satavaptan — tablets
  Other Names: SR121463
  Arms: Satavaptan Dose 1; Satavaptan Dose 2
Drug: placebo — tablets
  Arms: Placebo

SUMMARY:
The primary objective of this study is to assess the efficacy of satavaptan versus placebo in participants with dilutional hyponatremia due to SIADH.

Secondary objectives are to assess the safety of satavaptan, the maintenance of effect, and the clinical benefit in these participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants with symptomatic syndrome of inappropriate antidiuretic hormone secretion (SIADH) with chronic hyponatremia

Exclusion Criteria:

* Presence of clinical signs of hypovolemia (e.g. orthostatic decreases in blood pressure and increase in pulse rate, dry mucus membranes, decreased skin turgor)
* Presence of clinical signs of hypervolemia (e.g. generalized edema, jugular venous extension)
* Participants with adrenocortical insufficiency
* Participants with hypothyroidism
* Participants with known causes of transient SIADH
* Participants with psychogenic polydipsia or beer potomania
* Concomitant use of thiazide diuretics during the study
* Presence of uncontrolled diabetes with fasting blood glucose ≥200 mg/dL (≥11.09 mmol/L) at time of screening
* Participants with impaired hepatic function or liver cirrhosis (Child-Pugh A-C)
* Pregnant or breast-feeding women

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2008-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
serum sodium change from baseline | At Day 5 pre-dose

SECONDARY OUTCOMES:
responder rate | At Day 5 pre-dose
presence and intensity of clinical symptoms related to hyponatremia | At each scheduled visit
change from baseline in cognitive function | At Day 5 and 30

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States